CLINICAL TRIAL: NCT05052086
Title: Magnetomotoric Ultrasound (MMUS) in the Staging of Rectal Cancer
Brief Title: Magnetomotoric Ultrasound (MMUS) in Rectal Cancer
Acronym: MAMORECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MAMORECT
Record Dates: First submitted 2021-09-06; First posted 2021-09-22 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Included patients will undergo magnetomotoric ultrasound in addition to conventional MRI. The results of MRI examination and magnetomotoric ultrasound will be compared with final histopathology.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetomotoric ultrasound (Experimental): Magnetomotoric ultrasound in addition to MRI.
  Interventions: Diagnostic Test: Magnetomotoric ultrasound

INTERVENTIONS:
Diagnostic Test: Magnetomotoric ultrasound — Nanoparticles will be injected close to the tumor. Magnetomotoric ultrasound will be performed just before scheduled standard operation, when the patient is anesthetized.

SUMMARY:
Magnetomotoric ultrasound, combines conventional ultrasound with a time-varying magnetic field. The aim is to improve diagnosis of mesolectal lymph nodes.

DETAILED DESCRIPTION:
Magnetomotoric ultrasound, combines conventional ultrasound with a time-varying magnetic field. Nanoparticles are injected close to the rectal cancer and migrate to adjacent lymph nodes.The time-varying magnetic field will influence the nano particles in the lymph node enhancing diagnosis of affected lymph nodes. The aim is to improve diagnosis of mesolectal lymph nodes and compare the results of magnetomotoric ultrasound with MRI and final histopathology.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer
* Scheduled for total mesorectal surgery
* Informed consent

Exclusion Criteria:

* Not able to give informed consent
* Synchronus colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of mesorectal lymph node diagnosis with MMUS, compared with final histopathology | Approximately 1 hour after MMUS
  Evaluation of the accuracy of MMUS in detecting lymph node metastases in rectal cancer. The results of the MMUS (malignant or benign lymph nodes) will be compared with final histopathology. The accuracy will be expressed in sensitivity (%), specificity (%) and overall accuracy (% correctly staged lymph nodes with MMUS)
Accuracy of mesorectal lymph node diagnosis with MMUS, compared with preoperative MRI | Approximately 1 hour after MMUS
  Evaluation of the accuracy of MMUS in detecting lymph node metastases in rectal cancer in comparison to standard staging (MRI). The results of the MMUS (malignant nodes or benign nodes) will be compared with the results of preoperative MRI (malignant or benign lymph nodes) and the final histopathology. The accuracy will be expressed in sensitivity (%), specificity (%) and overall accuracy (% correctly staged lymph nodes) with MMUS and MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Skane University Hospital, Malmö, section of Surgery, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No